CLINICAL TRIAL: NCT05809830
Title: Phase I/II Randomized Trial of LB-100 Plus Doxorubicin vs. Doxorubicin Alone in First Line of Advanced Soft Tissue Sarcomas
Brief Title: Phase I/II of LB-100 Plus Doxorubicin vs. Doxorubicin Alone in First Line of Advanced Soft Tissue Sarcomas
Acronym: Enhancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-74
Record Dates: First submitted 2023-03-27; First posted 2023-04-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Advanced Soft-tissue Sarcoma
MeSH Terms: interventions — LB100; Doxorubicin

STUDY DESIGN:
Intervention Model Description: A Phase I dose-finding stage for the LB-100 plus doxorubicin combination is planned for an initial set of 9-18 patients (21-day cycles) In the Phase II part, patients will be enrolled in the trial via randomization. A randomization module (integrated in the eCRF system) will be used to assign patients to either the experimental arm (LB-100 plus doxorubicin) or to the control arm (doxorubicin alone) (1:1 ratio)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LB-100 plus doxorubicin (Experimental): * LB-100 will be administered during the first 3 days of each cycle (days 1, 2, and 3) at RP2D as a 2-hour intravenous infusion (with 500 mL of physiological saline solution), every 3 weeks (21-day cycles until progression or intolerance).
  * Doxorubicin will be administered only once (day 1) of each cycle at RP2D as a 20-minute infusion after completion of LB-100, every 3 weeks (up to a maximum of 6 x 21-day cycles).
  Interventions: Drug: LB-100 plus Doxorrubicin
- Doxorubicin alone (Active Comparator): Control: Doxorubicin will be administered only once (day 1) of each cycle at RP2D as a 20-minute infusion every 3 weeks (up to a maximum of 6 x 21-day cycles).
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: LB-100 plus Doxorrubicin — In Phase one the intervention will be LB-100 plus Doxorrubicin. The experimental arm in Phase II will also be LB-100 plus Doxorrubicin
  Arms: LB-100 plus doxorubicin
Drug: Doxorubicin — The control arm in Phase II will be Doxorrubicin alone
  Arms: Doxorubicin alone

SUMMARY:
A Phase I dose-finding stage for the LB-100 plus doxorubicin combination is planned for an initial set of 9-18 patients (21-day cycles). After that, in the Phase II part, patients will be randomized (ratio 1:1) to either the experimental arm (LB-100 plus doxorubicin combination) or the control arm (doxorubicin alone) to, comparatively, evaluate the efficacy of the LB-100 plus doxorubicin combination vs. doxorubicin alone

ELIGIBILITY:
Inclusion Criteria Phase I:

1. The patient must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging tests, etc.) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age ≥ 18 years.
3. Diagnosis of advanced/metastatic soft tissue sarcoma (undifferentiated pleomorphic sarcoma, leiomyosarcoma, myxoid and hypercellular myxoid liposarcoma, myxofibrosarcoma, NOS sarcoma, synovial sarcoma, fibrosarcoma, or malignant nerve sheath tumor) confirmed by central pathology review.
4. Mandatory pre-treatment formalin-fixed paraffin embedded (FFPE) tumor tissue must be provided for all subjects without exception for central pathology review and the translational study. If archive biopsy is not available or is older than 3 months, the patient must be willing to have a pre-treatment re-biopsy of primary or metastatic tumor (baseline biopsy) within 28 days prior to enrollment.
5. The patient must be willing to undergo a second mandatory biopsy just before the initiation of the 3rd cycle and agree that this sample is used for the translational study.
6. Measurable disease according to RECIST v1.1 criteria.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. The patient must be naïve of any previous treatment with anthracyclines (not even in adjuvant chemotherapy).
9. Adequate organ, hepatic, renal, cardiac, and hematologic function.
10. Laboratory tests as follows:

    * Absolute neutrophil count ≥ 1,200/mm³
    * Platelet count ≥ 100,000/mm³
    * Hg > 9 g/dL
    * Bilirubin ≤ 1.5 mg/dL
    * PT and INR ≤ 1.5
    * AST and ALT ≤ 2.5 times ULN
    * Creatinine ≤ 1.5 mg/dL or estimated creatinine clearance ≥ 60 mL/min
    * Blood glucose < 150 mg/dL
11. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan assessed within 28 days before enrollment.
12. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment. Patients must not be pregnant or nursing at study entry.
13. Women and men of reproductive potential must have agreed to use an effective contraceptive method during study treatment and for 3 months after the last dose of study drug.

Exclusion Criteria Phase I:

1. Diagnosis different from the elegible histological subtypes.
2. Previous treatment with doxorubicin, epirubicin, idarubicin, and/or other anthracyclines or any other systemic therapy. The exception is previous systemic therapy for a previous neoplasm (see exclusion criteria 10), if this is controlled, as long as it did not include anthracyclines.
3. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI CTCAE version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
4. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
5. Any of the following diseases/illnesses within the previous 6 months:

   * Myocardial infarction
   * Severe or unstable angina
   * Coronary or peripheral artery bypass graft
   * Cerebrovascular accident or transient ischemic attack (TIA)
   * Pulmonary embolism
6. Evidence of a bleeding diathesis.
7. Ongoing cardiac dysrhythmias > Grade 2.
8. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
9. History of allergy to study drug components.
10. History of another cancer with the exception of adequately treated basal cell carcinoma or in situ cervical cancer, or with a relapse-free interval longer than 3 years after treatment of the primary cancer with no substantial risk of recurrence.
11. Presence of brain or central nervous system metastases at the time of enrollment.
12. Patient is unwilling to provide mandatory translational tumor samples or biopsies (if required) cannot be easily taken.

Inclusion Criteria Phase II:

1. The patient must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging tests, etc.) and obtainedprior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age ≥ 18 years.
3. Diagnosis of advanced/metastatic soft tissue sarcoma (undifferentiated pleomorphic sarcoma or leiomyosarcoma) confirmed by central pathology review.
4. Mandatory pre-treatment formalin-fixed paraffin embedded (FFPE) tumor tissue must be provided for all subjects without exception for central pathology review and the translational study. If archive biopsy is not available or is older than 3 months, the patient must be willing to have a pre-treatment re-biopsy of primary or metastatic tumor (baseline biopsy) within 28 days prior to enrollment.
5. Measurable disease according to RECIST v1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. The patient must be naïve of any previous treatment with anthracyclines (not even in adjuvant chemotherapy).
8. Adequate organ, hepatic, renal, cardiac, and hematologic function.
9. Laboratory tests as follows:

   * Absolute neutrophil count ≥ 1,200/mm³
   * Platelet count ≥ 100,000/mm³
   * Hg > 9 g/dL
   * Bilirubin ≤ 1.5 mg/dL
   * PT and INR ≤ 1.5
   * AST and ALT ≤ 2.5 times ULN
   * Creatinine ≤ 1.5 mg/dL or estimated creatinine clearance ≥ 60 mL/min
   * Blood glucose < 150 mg/dL 10. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan assessed within 28 days before enrollment.

11. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment. Patients must not be pregnant or nursing at study entry.

12. Women and men of reproductive potential must have agreed to use an effective contraceptive method during study treatment and for 3 months after the last dose of study drug.

Exclusion criteria Phase II:

1. Diagnosis of any sarcoma different from undifferentiated pleomorphic sarcoma and leiomyosarcoma.
2. Previous treatment with doxorubicin, epirubicin, idarubicin, and/or other anthracyclines or any other systemic therapy. The exception is previous systemic therapy for a previous neoplasm (see exclusion criteria 10), if this is controlled, as long as it did not include anthracyclines.
3. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI CTCAE version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
4. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
5. Any of the following diseases/illnesses within the previous 6 months:

   * Myocardial infarction
   * Severe or unstable angina
   * Coronary or peripheral artery bypass graft
   * Cerebrovascular accident or transient ischemic attack (TIA)
   * Pulmonary embolism
6. Evidence of a bleeding diathesis.
7. Ongoing cardiac dysrhythmias > Grade 2.
8. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
9. History of allergy to study drug components.
10. History of another cancer with the exception of adequately treated basal cell carcinoma or in situ cervical cancer, or with a relapse-free interval longer than 3 years after treatment of the primary cancer with no substantial risk of recurrence.
11. Presence of brain or central nervous system metastases at the time of enrollment.
12. Patient is unwilling to provide mandatory translational tumor samples or biopsies (if required) cannot be easily taken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Maximun Tolerated Dose (MTD) (Phase I) | After six months
  The MTD of LB-100 in combination with doxorubicin will be determined by assessing adverse events according to CTCAE v5.0.
Progression-free survival (PFS) (Phase II) | After two years
  Efficacy measured by median PFS according to RECIST v1.1

SECONDARY OUTCOMES:
Adverse Events (Phase I and II) | Between six months and two years
  Safety profile/Toxicity assessed by adverse events related to study drugs
Overall Response Rate (ORR) (Phase I and II) | Between six months and two years
  Efficacy measured by the ORR, which is defined as the number of subjects with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) divided by the number of response evaluable subjects.
Progression-free survival (PFS) (Phase I) | After six months
  Efficacy measured by median PFS according to RECIST v1.1
Overall survival (OS) (Phase I and II) | Between six months and two years
  Censored on the last date a subject was known to be alive
EORTC QLQ-C30 questionnaire (Phase I and II) | Between six months and two years
  Quality of life assessed by using the EORTC QLQ-C30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín Broto, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz
Locations (6):
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No